CLINICAL TRIAL: NCT05156307
Title: Accuracy and Predictive Values for Colorectal Cancer of a Quantitative Faecal Immunochemical Test in Symptomatic Patients in Primary Care
Brief Title: Accuracy and Predictive Values for Colorectal Cancer of Quantitative FIT in Symptomatic Patients in Primary Care
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Region Örebro County (Other)
Collaborators: Region Jämtland Härjedalen (Other); Region Östergötland (Other); Uppsala County Council, Sweden (Other Government); Dalarna County Council, Sweden (Other); Landstinget i Värmland (Other)
Responsible Party: Principal Investigator, Louise Olsson, MD, PhD, Region Örebro County
Other Study IDs: 275691
Record Dates: First submitted 2021-12-01; First posted 2021-12-14 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-11

CONDITIONS: Colorectal Cancer
Keywords: Quantitative faecal immunochemical test, symptomatic, primary care
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to determine accuracy and predictive values for colorectal cancer of a faecal quantitative immunochemical test (FIT) in unselected symptomatic patients presenting in primary care. Main reference test will be linkage to a nationwide colorectal cancer registry.

DETAILED DESCRIPTION:
This is a nationwide multi-centre study in primary care, Sweden. Patients from the age of 40 years and above presenting in primary care with symptoms associated with colorectal cancer prompting their GP to take actions are eligible.

Consenting patients will fill out a short form on symptoms during last 4 weeks. They will provide 2 faecal samples from 2 different days. Samples will be analysed at any of three laboratories within 5 days using QuikRead go® (Aidian Oy). The analytical working range is 10-200 µg Hb/g faeces. The outcome will be reported as the concentration of first test (FIT 1) and highest concentration of two tests (FIT max). The outcome of the study FIT will remain within the study and GPs must request a separate FOBT for clinical purposes.

Reference test will be linkage to the Swedish Colorectal Cancer Registry (with in practice complete coverage) after at most 2 years for all patients. Accuracy and predictive values will be determined and ROC-curves analysed.

Some patients included in the study will be referred for colonoscopy for clinical reasons, and the outcome of FIT in relation to colonoscopy findings will be reported for this group as well.

ELIGIBILITY:
Inclusion Criteria:

Patients presenting in primary care with symptoms associated with colorectal cancer prompting their GP to take actions are eligible.

Exclusion Criteria:

Referral for bowel examination for other reasons than symptoms. Not able to understand the instructions for participation.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥ 40 years presenting in primary care with symptoms associated with colorectal cancer prompting their GP to take actions are eligible. This involves referral for any endoscopic or radiological examination of the large bowel, laboratory testing, including faecal occult blood test according to local routines, or clinical follow-up within soon. Both urgent referrals and patients planned for at least initial management in primary care are eligible, ie there will be no attempt to delimitate the study population based on any categorization of symptoms into "alarm" and "non-alarm" symptoms. The study population will be defined by primary care physicians´ clinical reasoning and assessment of colorectal cancer as a (more or less) possible diagnosis at the unique consultation.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Colorectal cancer | 2 years
  Linkage to cancer registry

CONTACTS AND LOCATIONS:
Overall Officials: Louise Olsson, MD, PhD, Principal Investigator — Region Örebro län, Camtö
Locations (1):
- Skebäcks VC, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Loov A, Hogberg C, Lilja M, Theodorsson E, Hellstrom P, Metsini A, Olsson L. Diagnostic accuracy for colorectal cancer of a quantitative faecal immunochemical test in symptomatic primary care patients: a study protocol. Diagn Progn Res. 2022 Aug 18;6(1):16. doi: 10.1186/s41512-022-00129-7. PMID 35978403